CLINICAL TRIAL: NCT05780918
Title: A Randomized Clinical Trial of Scenario Planning for Older Adults With Serious Injury
Brief Title: A Communication Tool to Improve Communication in the ICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Maryland, Baltimore (Other); University of California, Davis (Other); Harborview Injury Prevention and Research Center (Other); Lehigh Valley Health Network (Other); Grady Memorial Hospital (Other); Froedtert Hospital (Other); University of Alabama at Birmingham (Other); Rhode Island Hospital (Other); American College of Surgeons (Other); Coalition for National Trauma Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0334; R01AG078242-01 (NIH); Protocol Version 5/5/2025 (Other: UW Madison); A539750 (Other: UW Madison)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-05

CONDITIONS: Serious Injury; Communication
Keywords: intensive care unit; trauma; patient decision making; surgical decision making; shared decision making; decision support techniques
MeSH Terms: conditions — Communication; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial, sites randomized to start time.
  The intervention will be administered as a quality improvement activity because its primary purpose is to increase behaviors recommended by professional societies, e.g., timely communication with families and emotional support.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Case/Worst Case-ICU Communication Tool (Experimental): Patients in the intervention group will receive care from a trauma team that routinely uses the Best Case/Worst Case-ICU communication tool.
  Interventions: Other: Best Case/Worst Case-ICU Communication Tool
- Usual Care (No Intervention): Prior to implementation of the intervention, patients admitted to the trauma ICU will receive usual care. Usual care typically includes conversations focused on isolated problems, disarticulated from the patient's overall health trajectory. This is typified by the systems-base review, routinely summarizing each patient on rounds where the clinician lists each physiologic system, (e.g., neuro, cardiac, pulmonary…) with an assessment and plan to "fix" each abnormality with a new treatment. Deliberation about how these individual treatments align with patient preferences is typically prompted by major events like failure to liberate from a ventilator or imminent death. This pattern of usual care is well characterized and differs from daily scenario planning with the Best Case/Worst Case-ICU communication tool.

INTERVENTIONS:
Other: Best Case/Worst Case-ICU Communication Tool — This intervention uses scenario planning and a daily report of the interplay between major events and prognosis to illustrate a range of long-term outcomes and treatment experiences. By using a graphic aid to illustrate "what we are hoping for," "what we are worried about," and the evolution of the patient's story over time, the tool aims to facilitate dialogue among older adult trauma patients, their families, and the trauma team. Because the tool delivers critical prognostic information over the longitudinal course of care, subsequent treatment decisions can be made within the context of the patient's overall health status. This information alerts patients and families to the life-limiting nature of serious injury and provides an entrée for them to consider how comfort-focused strategies might better align with patients' end-of-life goals.
  All clinicians will be trained to create, use, and/or reference the graphic aids with patients depending on their roles in the trauma ICU.
  Arms: Best Case/Worst Case-ICU Communication Tool

SUMMARY:
The purpose of this study is to test the effectiveness of the Best Case/Worst Case-ICU communication tool on quality of communication, clinician moral distress, and ICU length of stay for older adults with serious traumatic injury. Investigators will follow an estimated 4500 patients aged 50 years and older who are in the ICU for 3 or more days and survey 1500 family members and up to 1600 clinicians from 8 sites nationwide.

DETAILED DESCRIPTION:
This is a multisite, stepped-wedge, randomized clinical trial. At the start of the study, investigators will randomly assign each site to the time when the intervention team will train all trauma surgeons, trainees, and ICU clinicians to use the Best Case/Worst Case-ICU tool. Participants in the intervention group will receive care from a trauma team that routinely uses the Best Case/Worst Case-ICU communication tool. Participants in the control group will receive usual care.

The study team will follow an estimated 4,500 patients with the highest post-injury mortality: aged 50 years and older with an ICU length of stay of 3 or more days. They will administer surveys to family members (quality of communication) and clinicians (moral distress) and obtain patient-level outcomes (ICU length of stay (LOS)), clinical data, and demographics from the Trauma Quality Improvement Program (TQIP) national registry.

Objectives:

* Aim 1: To test the effectiveness of the Best Case/Worst Case-ICU communication tool on improving the quality of communication in the trauma ICU.
* Aim 2: To test the effectiveness of the Best Case/Worst Case-ICU communication tool on reducing clinician moral distress in the ICU.
* Aim 3: To test the effectiveness of the Best Case/Worst Case-ICU communication tool on reducing ICU length of stay.

ELIGIBILITY:
Patients

Inclusion Criteria:

* aged 50 and older
* admitted to the ICU for 3 or more days after serious injury

Exclusion Criteria:

* none

Family Members

Inclusion Criteria:

* aged 18 and older
* patient's family member or informally designated "like family" or primary surrogate decision maker
* speak English or Spanish

Exclusion Criteria:

* does not have decision-making capacity

Clinicians

Inclusion Criteria:

* provide care in the trauma ICU (including attending trauma surgeons, fellows, residents, advance practice providers, bedside nurses and medical assistants, respiratory techs and physical therapists, social workers, and chaplains)

Exclusion Criteria:

* do not provide care in the trauma ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7600 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Family-reported Quality of Communication (QOC) within 5-7 days of ICU admission | up to 10 days after patient admission, one-time survey for family members
  Family-reported quality of communication will be measured using the 20-item Quality of Communication (QOC) scale. The QOC is a validated self-report instrument. The average composite score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.

SECONDARY OUTCOMES:
Family-reported General Quality of Communication (QOC), within 5-7 days of ICU admission | up to 10 days after patient admission, one-time survey for family members
  Family-reported general quality of communication will be measured using the 6-item general communication subscale of the 20-item quality of communication (QOC) scale. The QOC is a validated self-report instrument. The average item score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.
Family-reported End-of-Life (EOL) Quality of Communication (QOC), within 5-7 days of ICU admission | up to 10 days after patient admission, one-time survey for family members
  Family-reported quality of end-of-life communication will be measured using 7-item end-of-life communication subscale of the 20-item Quality of Communication scale. The QOC is a validated self-report instrument. The average item score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.
Family-reported proportion of Goal Concordant Care (GCC) at 5-7 days post ICU admission | up to 10 days after patient admission, one-time survey for family members
  Family-reported goal-concordant care will be assessed by 2 survey questions taken from the SUPPORT study. (Question 1 - Preferences for Care: If you had to make a choice at this time, would you prefer a course of treatment for your loved one that focuses on extending life as much as possible, even if it means having more pain and discomfort, or would you want a plan of care that focuses on relieving pain and discomfort as much as possible, even if that means not living as long? Question 2 - Current Receipt of Care Consistent With Preferences: Would you say that your loved one's current medical care is more focused on extending life as much as possible, even if it means having more pain and discomfort, or on relieving pain and discomfort as much as possible, even if that means not living as long?) If participant gives the same answer to both questions, this will be considered concordant. If the answers to the two questions are different, this will be considered discordant.
Clinician-reported Measure of Moral Distress for Healthcare Professionals (MMD-HP) | 3 months prior to each implementation wave and again 12 months later
  As a proximate measure of the intervention effect on ICU conflict, the investigators will use the Measure of Moral Distress for Health Care Professionals (MMD-HP) to measure center-level distress at the beginning and the end of the study. Frequency and level of distress of clinician experiences are each rated on a 0-4 scale where 0 is 'never' and 4 is 'very frequently' and 0 is 'none' and 4 is 'very distressing,' respectively. The total possible range of scores is 0-432 (the product of the frequency times the level of distress for 27 items) with higher scores indicating more moral distress.
Clinician-reported Emotional Exhaustion (EE) - Maslach Burnout Inventory (MBI) | 3 months prior to each implementation wave and again 12 months later
  Clinician emotional exhaustion will be measured with the Maslach Burnout Inventory - Human Services Survey (MBI-HSS), a 22-item inventory scored on a 7 point Likert scale from 0-6 where 0 is 'never' and 6 is 'everyday'. The EE subscale includes 9 items for a total possible range of scores from 0-54, higher scores indicate increased emotional exhaustion.
Clinician-reported Depersonalization (DP) - Maslach Burnout Inventory (MBI) | 3 months prior to each implementation wave and again 12 months later
  Clinician depersonalization will be measured with the Maslach Burnout Inventory - Human Services Survey (MBI-HSS), a 22-item inventory scored on a 7 point Likert scale from 0-6 where 0 is 'never' and 6 is 'everyday'. The DP subscale includes 5 items for a total possible range of scores from 0-30, higher scores indicate increased depersonalization.
Clinician-reported Personal Accomplishment (PA) - Maslach Burnout Inventory (MBI) | 3 months prior to each implementation wave and again 12 months later
  Clinician personal accomplishment will be measured with the Maslach Burnout Inventory - Human Services Survey (MBI-HSS), a 22-item inventory scored on a 7 point Likert scale from 0-6 where 0 is 'never' and 6 is 'everyday'. The PA subscale includes 8 items for a total possible range of scores from 0-48, higher scores indicate decreased personal accomplishment.
Patient ICU Length of Stay (LOS) | during hospitalization, provided by TQIP at study completion (estimated up to 2 years)
  ICU LOS will be measured as the cumulative amount of time each study qualified patient spent in the ICU during the post-injury hospital admission. Each partial or full day is measured as one calendar day.
Patient Total Time on Ventilator | during hospitalization, provided by TQIP at study completion (estimated up to 2 years)
  Patient total time on ventilator will be measured as the cumulative amount of time each study qualified patient spent on a ventilator during the post-injury hospital admission. Each partial or full day is measured as one calendar day.
Patient Time to In-hospital Death | during hospitalization, provided by TQIP at study completion (estimated up to 2 years)
  Dichotomous variable (alive or deceased) at hospital discharge
Patient 6-month Mortality | 6 months after patient admission, provided by TQIP at study completion (estimated up to 2 years)
  The procedure for death ascertainment at 6 months after admission includes chart review, attempt to reach listed patient contacts, and internet search. Patients without documentation of death will be presumed alive. Dichotomous variable (presumed alive or confirmed deceased).
Patient Time to Withdrawal of Life Supporting Treatment | during hospitalization, provided by TQIP at study completion (estimated up to 2 years)
  Withdrawal of life-supporting treatment will be measured as the cumulative amount of time between each study qualified patients' admission and withdrawal of life supporting treatment at the end of life. Each partial or full day is measured as one calendar day.

OTHER OUTCOMES:
Practitioner Opinion Survey | at study completion (estimated up to 2 years)
  To evaluate the implementation of the intervention, trauma surgeons will be asked for their impressions of the Best Case/Worst Case-ICU communication tool using a 12-item questionnaire upon study completion. Each question is measured on an ordinal, 5-point Likert scale where 1 is 'strongly disagree' and 5 is 'strongly agree.'

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Schwarze, MD, MPP, Principal Investigator — University of Wisconsin, Madison
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis Medical Center, Davis, California
  - Grady Memorial Hospital - Morehouse School of Medicine, Atlanta, Georgia
  - Shock Trauma - University of Maryland Medical Center, Baltimore, Maryland
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Rhode Island Hospital - Brown University, Providence, Rhode Island
  - Harborview Medical Center - University of Washington, Seattle, Washington
  - Froedtert Hospital - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set comprised of survey data, metadata, and analytic code will be made available through the National Archive of Computerized Data on Aging (NACDA) or comparable NIH-supported repository. A de-identified data set describing the implementation of the intervention will also be made available, including dates of cross-over into the intervention arm, training dates, notes from training sessions, and a data supplement that includes general information about the project that will provide context of the data. This will include a final study protocol, data dictionary, information sheets, and copies of all survey data collection tools.
  Patient-level data used for this project, originally collected by the Trauma Quality Improvement Program (TQIP) Registry, will not be made available for sharing by the University of Wisconsin. This data is available upon request from the American College of Surgeons (ACS), who administer the TQIP program.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All de-identified data will be made available within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: Data housed in NACDA or comparable NIH-supported repository will be restricted and researchers seeking access must complete a Restricted Data Use Agreement required by the repository, including documenting how regulatory requirements at their institution have been met and providing a data security plan. Once the repository receives and approves the agreement, repository staff will send the requestor an encrypted link to obtain the data files.

REFERENCES:
- [Derived] Stalter L, Hanlon BM, Bushaw KJ, Kwekkeboom KL, Zelenski A, Fritz M, Buffington A, Stein DM, Cocanour CS, Robles AJ, Jansen J, Brasel K, O'Connell KM, Cipolle MD, Ayoung-Chee P, Morris R, Gelbard RB, Kozar RA, Lueckel S, Schwarze M. Best Case/Worst Case-ICU: protocol for a multisite, stepped-wedge, randomised clinical trial of scenario planning to improve communication in the ICU in US trauma centres for older adults with serious injury. BMJ Open. 2024 Aug 28;14(8):e083603. doi: 10.1136/bmjopen-2023-083603. PMID 39209498